CLINICAL TRIAL: NCT06220097
Title: Study on the Safety and Efficacy of Mitoxantrone Hydrochloride Liposome Injection-containing Bridging Regimen in CD19-targeting CAR-T Therapies
Brief Title: Mitoxantrone Hydrochloride Liposome Injection-containing Bridging Regimen and CD19-targeting CAR-T Therapies
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Collaborators: CSPC Pharmaceutical Group Limited (Industry)
Responsible Party: Principal Investigator, MEI HENG, : Proferssor, Cheif Doctor, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: bridging regimen of CD19CAR-T
Record Dates: First submitted 2024-01-11; First posted 2024-01-23 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-01

CONDITIONS: B-cell Acute Lymphoblastic Leukemia; B-cell Lymphoma Refractory
MeSH Terms: conditions — Burkitt Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Effective of MHL injection-containing bridging regimens with CD19 CAR-T (Experimental): After enrollment, all subjects will receive a combination regimen of mitoxantrone hydrochloride liposomal injection within 28 days to 7 days before CAR-T infusions will be included, including but not limited to the R-MINE regimen (mitoxantrone hydrochloride liposomal injection combined with rituximab, mesna, ifosfamide and etoposide), G-MINE regimen (mitoxantrone hydrochloride liposomal injection combined with obinutuzumab, mesna, ifosfamide and etoposide), MAE scheme (mitoxantrone hydrochloride liposomal injection combined with cytarabine, etoposide), etc.
  Interventions: Drug: Mitoxantrone hydrochloride liposome Injection-based bridging therapy+ Fludarabine-based chemotherapy +CD19 CAR-T Cells

INTERVENTIONS:
Drug: Mitoxantrone hydrochloride liposome Injection-based bridging therapy+ Fludarabine-based chemotherapy +CD19 CAR-T Cells — Bridging therapies from enrollment before CD19 CAR-T infusion. A treatment regimen containing mitoxantrone hydrochloride liposome injection, including but not limited to the following recommended regimens: R-MINE regimen (rituximab + ifosfamide + mitoxantrone hydrochloride liposome + etoposide) G-MINE regimen (obinutuzumab + ifosfamide + mitoxantrone hydrochloride liposome + etoposide) MAE regimen (mitoxantrone liposome hydrochloride + cytarabine + etoposide) . The recommended dose of mitoxantrone liposome hydrochloride is not limited. For patients who achieve SD or better after one cycle of bridging treatment, it is up to the investigator to decide whether to receive CAR-T therapy. Fludarabine-based lymphodepletion chemotherapy was followed by CD19 CAR-T cells (relma-cel, axi-cel or humanized CAR19). Relma-cel and axi-cel will be infused according to the instructions. CART19 infusion is conducted at a dose of 1x10^6/kg on day 0 and day 1 respectively.

SUMMARY:
The goal of this open, single-arm practical, phase II, clinical study is to evaluate the efficacy and safety of the mitoxantrone hydrochloride liposome injection-containing regimens in bridging therapies of CD19 CAR-T cells. The main question it aims to answer is:

• the efficacy of the mitoxantrone hydrochloride liposome injection-containing combination regimens in bridging therapies of CD19 CAR-T cells.

Participants will receive combination bridging regimens including mitoxantrone hydrochloride liposomal injection and CAR-T cell therapy to see if the combination regimens have a positive effect on the efficacy of bridging therapies.

DETAILED DESCRIPTION:
Chimeric antigen receptor T-cell (CAR-T) therapy has been approved for a variety of relapsed/refractory hematologic malignancies and has significantly improved patient outcomes. The preparation of CAR-T cells, including a variety of relevant individual factors, usually takes at least 3-4 weeks, or more, so patients may require bridging therapy (BT) to control disease progression and prevent the rapid exacerbation of systemic cancer. Clinical trial data have shown that about 7% of patients do not survive while waiting for CAR-T cell preparation to be completed, so individual bridging therapy can be given after apheresis and 4-6 weeks before CAR-T infusion to achieve effective CAR-T cell therapy.

Mitoxantrone, a traditional anthracycline quinone, is an antibiotic antineoplastic drug. It exerts antitumor effects by interfering with DNA, RNA, and inhibition of topoisomerase II, and is a cell cycle non-specific drug[]. Liposomes are excellent carriers of anti-tumor drugs, which can reduce the distribution of drugs in normal tissues and increase the accumulation of drugs in tumor tissues, thereby reducing toxicity and improving treatment efficacy. To reduce the toxicity of mitoxantrone and improve its efficacy, CSPC Pharmaceutical Group has developed the liposomal formulation of mitoxantrone, which is based on liposomal R&D technology. A new technical upgrade has been carried out on the mitoxantrone liposome, making it the only liposome with a higher dosage than the ordinary preparation, and it is a new anthracycline liposome that has been comprehensively upgraded. In the pivotal phase II study of liposomal mitoxantrone, monotherapy with PTCL was associated with an ORR of 41.7%, a CR rate of 23.1%, a median PFS of 8.5 months, a median OS not reached, and a high incidence of adverse events such as neutropenia and pigmentation, with a good cardiac safety profile and no progression of cardiotoxicity. Single-agent 16mg/m2 and 20mg/m2 doses were also explored in DLBCL, and 35 patients with relapsed and refractory DLBCL were enrolled, with an overall objective response rate of 38.5% in the 26 full analysis sets, which had certain activity in DLBCL.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥ 18 years and <75 years.
2. Eastern Cooperative Oncology Group score≤ 2.
3. Clinically diagnosed refractory or relapsed B-cell malignancies. Relapse refers to "relapse after a complete response (CR) from initial chemotherapy"; refractory refers to "diagnosis can be made if any of the following are met:(1) tumor shrinkage of <50% or disease progression (PD) after standard chemotherapy; (2) CR is achieved by standard chemotherapy but relapses within six months, (3) 2 or more recurrences after CR, (4) recurrence after hematopoietic stem cell transplantation"; B-cell malignancies include the following 3 categories: (1) B-cell acute lymphoblastic leukemia (B-ALL); (2) indolent B-cell lymphoma (CLL, FL, MZL); (3) aggressive B-cell lymphoma (DLBCL, BL, MCL).
4. Flow cytometry (FCM) or immunohistochemistry showed positive CD19 expression in tumor cells;
5. Organ function needs to meet the following conditions:

1) EF >50%, and there is no obvious abnormality on ECG; 2) SpO2≥90%； 3) Cr≤2.5 ULN; 4) ALT and AST≤5 ULN, TBil≤3 ULN; 6. Negativity of blood pregnancy test for women, and participants use effective methods of contraception until the last follow-up. 7. The patient or his or her legal guardian voluntarily participates in and signs an informed consent form.

Exclusion Criteria:

1. Prior treatment with doxorubicin or other anthracyclines with a total cumulative dose of doxorubicin >360 mg/m2 (other anthracyclines convert 1 mg of doxorubicin to 2 mg epirubicin).
2. Hypersensitivity to any of the study drugs or their components.
3. Concomitant other diseases that are not effectively controlled, including but not limited to persistent or poorly controlled infections, symptomatic congestive heart failure, unstable angina, cardiac arrhythmias, poorly controlled pulmonary diseases, or psychiatric disorders.
4. Investigators judge patients with central nervous system involvement who may be at high risk of receiving bridging therapy and CD19 CAR-T cell treatment.
5. Participants with other active malignancies within five years.
6. Patients with relapse after allogeneic hematopoietic stem cell transplantation who have had grade 3~4 acute graft-versus-host response (GVHD).
7. Patients who are pregnant or breast-feeding.
8. Active autoimmune disease requiring systemic immunosuppressive therapy.
9. Other conditions considered to increase the risk to the subject or interfere with the results of the trial by the researcher.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
The overall response rate (ORR) of patients after bridging therapy | After bridging therapy and before CD19 CAR-T infusion
  The overall response rate (ORR) was based on the Lugano 2014 Lymphoma Efficacy Evaluation Criteria (Cheson 2014) and the 2021 version of the ALL Efficacy Evaluation Index

SECONDARY OUTCOMES:
Complete response rate (CR) of patients after bridging therapy and CD19 CAR-T infusion | within 2 years after infusion
  CR will be assessed from CAR-T cell infusion to death or last follow-up (censored)
In vivo expansion and survival of CD19 CAR-T cells | within 2 years after infusion
  The quantity of CD19 CAR copies in bone marrow, peripheral blood and cerebrospinal fluid will be determined by using a quantitative polymerase chain reaction.
Incidence of Treatment-related Adverse Events | before bridging therapy and within 2 years after infusion
  Therapy-related adverse events (AE), including severe adverse events (SAE) and laboratory outliers with clinical significance, will be recorded and assessed according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE, Version 5.0).

CONTACTS AND LOCATIONS:
Locations (1):
- Union Hospital, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No